CLINICAL TRIAL: NCT05620524
Title: Therapeutic Oncolytic Monitoring as a Tool for Effective Exposure to 5-FU in Patients With Locally Advanced, Resectable Gastric or Gastro-oesophageal Junction Cancer Treated With Perioperative FLOT
Acronym: THOMAS FU FLOT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Thomas Manten, MSc., Catharina Ziekenhuis Eindhoven
Other Study IDs: THOMAS FU FLOT-001
Record Dates: First submitted 2022-11-10; First posted 2022-11-17 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: TDM of 5-FU; Pharmacokinetic Observational Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients treated with FLOT regimen: Exposure to 5-FU in patients treated with FLOT
  Interventions: Drug: Extra blood samples for determining exposure to 5-FU

INTERVENTIONS:
Drug: Extra blood samples for determining exposure to 5-FU — Extra blood samples for determining exposure to 5-FU

SUMMARY:
Traditional dosing of 5-FU is based on body surface area and DPD enzyme activity. However, BSA-based dosing is associated with wide inter-individual variations in 5-FU systemic exposure, and also 5-FU-induced toxicity. The international association for therapeutic drug monitoring and clinical toxicology (IATDMCT) state in there clinical guideline, in which all previous clinical pharmacokinetic studies of 5-FU were reviewed, that only 25% of the patients are within the therapeutic range. In the traditional treatment regimens a bolus of 400 mg/ m2 5-FU is given, followed by a dose of 2400 mg/m2 as a 46-hour infusion. The therapeutic range of 5-FU in these older regimens is defined by a target AUC of 20-30 mg*h/L. In contrast, 5-FU in FLOT regimen is given without a bolus, and in a high dose of 2600 mg/m2 as a 24-hour infusion. This means that a comparable absolute dose of 5-FU is given with FLOT and the older regimens, however, the manner and duration of administration differ. Based on this administration, it is expected that the FLOT regimen will result in an approximately two-fold higher steady state concentration (Css), as it is given in an approximately two-fold shorter period of time (t). As a result of this pharmacokinetic predictions, the exposure to 5-FU (AUC = Css x t) will be comparable between these different 5-FU regimens. Therefore, we hypothesise that the therapeutic range of 5-FU in FLOT will be comparable to the target AUC of 20-30 mg*h/L in the older regimens. Similar to the older treatment regimens, we expect that a significant part of patients will be outside this therapeutic window. To test these hypotheses, the aim of this study is to establish the population exposure of 5-FU in FLOT treatment regimen, and to determine the percentage of patients that achieves this therapeutic range.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed malignancy for which treatment with 5-FU is indicated in the FLOT regimen.
2. Age ≥ 18 years
3. Patient is able and willing to give written informed consent
4. WHO performance status 0-2
5. Patient fulfills the general treatment criteria for treatment with FLOT including appropriate liver and renal function and other standard applicable laboratory values
6. Patient is able and willing to undergo extra blood sampling for 5-FU analysis

Exclusion Criteria:

1. Patients with known substance abuse, psychotic disorders, and/or other diseases expected to interfere with study or the patient's safety.
2. Inability to undergo additional blood sampling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced, resectable gastric or gastro-esophageal junction cancer treated with perioperative FLOT.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-12-19 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Population exposure to 5-FU | 1 year
  AUC of 5-FU in FLOT treated patients

CONTACTS AND LOCATIONS:
Locations (1):
- Catharina hospital, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No